CLINICAL TRIAL: NCT02757105
Title: Randomized, Double-blind, Placebo-controlled, Phase 2 Trial of BEKINDA (Ondansetron 12 mg Bimodal Release Tablets) for Diarrhea Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of BEKINDA (Ondansetron 12 mg Bimodal Release Tablets) for Diarrhea Predominant Irritable Bowel Syndrome (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHB-102-02
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): BEKINDA 12 mg (Ondansetron Bimodal Release Tablets), once daily for 8 weeks
  Interventions: Drug: BEKINDA
- Group B (Placebo Comparator): Placebo, once daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BEKINDA
  Other Names: RHB-102 12 mg; Ondansetron Bimodal Release Tablet 12 mg
  Arms: Group A
Drug: Placebo
  Arms: Group B

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-arm parallel group study. After qualifying for the study and signing informed consent, patients will undergo a two-week observation period during which stool consistency and frequency data and symptom data will be collected. Patients will then be randomized 60:40 to RHB-102 12 mg (BEKINDA) or placebo. Patients will continue on treatment for 8 weeks. Each medication will be given once daily.

DETAILED DESCRIPTION:
All patients will undergo baseline evaluation including full history and physical, with particular attention to gastrointestinal symptomatology and findings, a standard set of safety laboratory examinations (CBC and platelet count, biochemical profile, urinalysis, serum thyroid-stimulating hormone (TSH) and free T4, INR), and 12-lead ECG. In addition, the following studies will be performed to exclude other causes of gastrointestinal symptoms:

* Serum testing for C-reactive protein and gluten sensitivity
* Colonoscopy if required per protocol
* Patients with a history of positive tests for ova, parasites or Clostridium difficile must undergo repeat testing, which must be negative, during the screening period. Starting during the baseline observation phase, all patients will keep diaries of symptomatology and stool frequency and consistency. Stool consistency will be assessed according to the Bristol Stool Form scale (Lewis and Heaton, 1997).

Patients will keep diaries of stool frequency and consistency, symptoms, study medication compliance, and use of all medications, including rescue medications, throughout the study.

Serum electrolyte assays (bicarbonate, calcium, chloride, magnesium, potassium, and sodium) will be performed at week 3 on study. Safety laboratory examinations will be performed during and after the treatment period in accordance with the study procedures schedule below.

Patients will be questioned periodically regarding concomitant medication use and the occurrence of adverse events.

Patients must complete at least 12 days of all baseline diary entries within the 14 day screening period to be eligible to participate in the study. Patients completing fewer than 12 days of diary entries may, at the investigator's discretion, repeat the screening period diary. As long as the patent can complete and enter the study within 6 weeks, baseline laboratory studies need not be repeated. If repeating the 2 weeks' baseline diary will result in a period longer than 6 weeks from consent to start of treatment, the medical monitor must be consulted prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age≥18 years (with a minimum of 35% males in the study)
2. Patient meets FDA guidance and Rome III criteria for IBS-D:

   a. Recurrent abdominal pain or discomfort over ≥6 months, with frequency ≥3 days/month in the last 3 months associated with ≥2 of the following: i. Improvement with defecation ii. Onset associated with a change in frequency of stool iii. Onset associated with a change in the form of stool b. Loose or watery stools (Bristol stool form scale 6 or 7) ≥2 days per week
3. Average worst daily pain intensity ≥3.0 for each of the two baseline weeks
4. Major laboratory parameters within the following limits (no worse than grade 1 abnormalities per NCI-CTCAE v4):

   a. Adequate hematologic function, as demonstrated by i. Hemoglobin ≥10 g/dL ii. Absolute neutrophil count (ANC) 1.5-10 x 10^9/L iii. Platelets ≥100 x 10^9/L b. Adequate liver and renal function as demonstrated by i. Aspartate transaminase (AST) and Alanine transaminase (ALT) each ≤ 3.0 x upper limit of normal (ULN) ii. Total bilirubin ≤1.5 x ULN iii. Creatinine ≤1.5 X ULN c. Euthyroid based on thyroid-stimulating hormone (TSH) and free T4 levels
5. Patients on thyroid hormone replacement must be on a stable dose for at least one month prior to study entry.
6. C-reactive protein ≤2 x ULN for lab
7. Patients of childbearing potential and male patients with partners of childbearing potential must utilize effective contraceptive measures Women of childbearing potential are women who have menstruated in the past 12 months, with the exception of women who have undergone surgical sterilization
8. All patients must sign informed consent.

Exclusion Criteria:

1. Evidence of other cause for bowel disease:

   1. Relevant abnormalities seen on colonoscopy if previously performed or if required per this protocol. These include but are not limited to Crohn's disease, ulcerative colitis, diverticulitis, ischemic colitis, microscopic colitis.
   2. History of and/or positive serologic test for celiac disease
   3. Known or suspected lactose intolerance.
2. History of abdominal surgery other than appendectomy or cholecystectomy at any time
3. Any elective major surgery (of any organ) planned for the period of the study, including follow-up
4. History of organic abnormalities of the GI tract including but not limited to intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, adhesions or impaired intestinal circulation (e.g., aortoiliac disease)
5. Current or previous diagnosis of neoplasia (except non-GI neoplasia in complete remission ≥5 years, squamous and basal cell carcinomas). With approval of the medical monitor patients with curatively treated neoplasm in complete remission <5 years may be entered in the study.
6. Patients with a history of positive tests for ova or parasites or Clostridium difficile must be retested during the screening period and tests for the relevant agents must be negative
7. Use of any 5-HT3 antagonist (5hydroxytryptamine receptor antagonists) within 4 weeks of the start of baseline data collection.
8. Use of rifaximin within 4 months of the start of baseline data collection.
9. Use of any other agent specific for IBS (such as alosetron or eluxadoline) or for symptomatic treatment of IBS (such as antispasmotics and antidiarrheals other than loperamide) within 2 weeks of the start of baseline data collection.
10. Uses of any investigational agent for any indication within 4 weeks of the start of baseline data collection.
11. Congestive heart failure, bradyarrhythmia (baseline pulse<55/min), known long QT syndrome
12. Patients who have Corrected QT interval (QTc) prolongation>450 msec noted on screening ECG, or who are taking medication known to cause QT prolongation

    Note: For current list of medications known to cause QT prolongation see:

    https://www.crediblemeds.org/healthcare-providers/drug-list/ There are several risk categories. Use the list showing those drugs known to cause torsade de pointes (TdP)
13. Hypersensitivity or other known intolerance to ondansetron or other 5-HT3 antagonists
14. Patient has taken apomorphine within 24 hours of screening
15. Pregnant or lactating
16. Patients with other major illnesses, either physical or psychiatric, or social situations which may interfere with participation in the study or interpretation of results
17. Patients with severe hepatic impairment, defined as Child-Pugh score ≥10 at baseline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - E Squared Research, Inc., Huntsville, Alabama
  - Endoscoopy Center of AR, Little Rock, Arkansas
  - Arkansas Gastroenterology, P.A., North Little Rock, Arkansas
  - Prx Clinical, Garden Grove, California
  - Providence Clinical Research, North Hollywood, California
  - Shahram Jacobs MD, Inc., Sherman Oaks, California
  - Advanced Rx Clinical Research Group, Inc., Westminster, California
  - Bristol Hospital Dba Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Clinical Research of Homestead, Homestead, Florida
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Great Lakes Medical Research, Mentor, Ohio
  - Clinsearch, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Aztec Medical Research, LLC, Channelview, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RHB-102: 1 tablet containing 3 mg immediate release and 9 mg sustained release ondansetron, once daily for 8 weeks
- Placebo: 1 tablet of matching placebo, once daily for 8 weeks
Period: Overall Study
Arm/Group | RHB-102 | Placebo
Started | 75 | 52
Treated (1 patient in the placebo group was randomized and not treated.) | 75 | 51
Completed (At least 7.6 weeks of treatment & end of study visit 28 +/- 11 days after last intake of study drug.) | 63 | 41
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RHB-102 | Placebo | Total
Number analyzed (Participants) | 75 | 51 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 49 | 120
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 35 | 88
  Male | 22 | 16 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 11 | 6 | 17
  Black or African American | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 58 | 42 | 100
  Other | 1 | 0 | 1
  Hispanic/Latino | 9 | 4 | 13
  Not Hispanic/Latino | 66 | 47 | 113
Median C-reactive protein (CRP) [Number; unit: mg/L] | 2.07 | 2.25 | 2.09

OUTCOME MEASURES:

1. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate - mITT Population
Description: A weekly stool consistency responder was defined in the FDA guidance on IBS-D as a patient who experienced (during a week) a ≥50% reduction in the number of days with at least one stool that has a consistency of Type 6 or 7 on the Bristol stool scale compared with baseline. In addition, to be considered a responder for the week, the patient could not have had an increase in average abdominal pain >10% over baseline during that week. A patient was characterized as an overall stool consistency responder if the patient was a weekly responder for at least 50% of the planned weeks of treatment.
Time Frame: 8 weeks
Population: Modified intent-to-treat (mITT) population analyzed included all patients who took at least one dose of double blinded study drug after randomization. In the mITT population, patients were analyzed by the treatment to which they were randomized. The population was used for a statistical analysis of efficacy endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 75 | 51
Participants
  Response | 42 | 18
  Non-response | 33 | 33
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.036, Chi-squared, Corrected

2. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate Males - mITT Population
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 22 | 16
Participants
  Response | 11 | 5
  Non-response | 11 | 11
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.410, Chi-squared, Corrected

3. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate Females - mITT Population
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 1 tablet matching placebo, once daily for 8 weeks
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 53 | 35
Participants
  Response | 31 | 13
  Non-response | 22 | 22
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.081, Chi-squared, Corrected

4. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate: Sensitivity Analysis Without Imputation for Use of Rescue Medication - mITT Population
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 75 | 51
Participants
  Response | 43 | 19
  Non-response | 32 | 32
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.042, Chi-squared, Corrected

5. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate by Baseline CRP > Median - mITT Population
Description: as for outcome 1
Time Frame: 8 weeks
Population: Patients with Baseline CRP > Median
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 37 | 26
Participants
  Response | 22 | 6
  Non-response | 15 | 20
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.009, Chi-squared, Corrected

6. Primary Outcome: Summary and Analysis of Overall Stool Consistency Response Rate by Baseline CRP ≤ Median - mITT Population
Description: as for outcome 1
Time Frame: 8 weeks
Population: Patients with Baseline CRP ≤ Median
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 38 | 25
Participants
  Response | 20 | 12
  Non-response | 18 | 13
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.919, Chi-squared, Corrected

7. Secondary Outcome: Summary and Analysis of Overall Worst Abdominal Pain Response Rate - mITT Population
Description: A weekly pain responder was defined as a patient who experienced a decrease in the weekly average of worst abdominal pain in the past 24 hours score ≥30% compared with baseline and no increase in the number of days per week with Type 6 or 7 stool consistency. An overall pain responder was defined as a patient who was a weekly pain responder for at least 50% of the planned weeks of treatment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 75 | 51
Participants
  Response | 38 | 20
  Non-response | 37 | 31
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.278, Chi-squared, Corrected; Mean Difference (Final Values) = 11.5, 95% CI 2-sided [-7.7 to 30.6]

8. Secondary Outcome: Summary and Analysis of Overall Study Response Rate - mITT Population
Description: A patient was characterized as an overall weekly responder if the patient met both the stool consistency and pain response definitions for a given week. A patient was characterized as a composite study responder if the patient met the criteria for both weekly stool consistency and pain response for at least 50% of the planned weeks of treatment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo
Number analyzed (Participants) | 75 | 51
Participants
  Response | 30 | 13
  Non-response | 45 | 38
Statistical Analysis 1: Comparison: RHB-102 vs Placebo; Test type: Superiority; p = 0.135, Chi-squared, Corrected; Mean Difference (Final Values) = 14.5, 95% CI 2-sided [-3.4 to 32.5]

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | RHB-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/51
Other Adverse Events (participants affected / at risk) | 68/75 | 47/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-102 (N=75) | Placebo (N=51)
Constipation TEAE (Gastrointestinal disorders) | 10 | 2
Flatulence TEAE (Gastrointestinal disorders) | 6 | 0
Urinary Tract Infection TEAE (Infections and infestations) | 4 | 1
Alanine aminotransferase increased TEAE (Investigations) | 6 | 2
Aspartate aminotransferase increased TEAE (Investigations) | 6 | 5
Blood creatinine increased TEAE (Investigations) | 5 | 2
Blood glucose increased TEAE (Investigations) | 17 | 9
Blood magnesium increased TEAE (Investigations) | 5 | 2
Blood potassium increased TEAE (Investigations) | 5 | 2
Blood sodium decreased TEAE (Investigations) | 4 | 7
Hemoglobin decreased TEAE (Investigations) | 5 | 3
Lymphocyte count decreased TEAE (Investigations) | 5 | 5
Protein urine present TEAE (Investigations) | 27 | 17
White blood cells urine positive TEAE (Investigations) | 23 | 17
pH urine increased TEAE (Investigations) | 4 | 1
Headache TEAE (Nervous system disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agree that the Sponsor shall have the right to the first publication of the results of the Study. Following the first publication, the PI may publish data or results from the Study; subject to Sponsor for review and approval in writing at least sixty (60) days prior to the date of the publication. Sponsor may require changes and may extend the embargo to protect its intellectual property or other proprietary interests and to allow for the taking actions for this purpose.

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT02757105/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02757105/SAP_001.pdf